CLINICAL TRIAL: NCT01517997
Title: Infrapopliteal Drug Eluting Angioplasty Versus Stenting for the Treatment of Long-segment Arterial Disease: The IDEAS-I Randomized Controlled Trial.
Brief Title: Infrapopliteal Drug Eluting Angioplasty Versus Stenting
Acronym: IDEAS-I
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, SIABLIS DIMITRIOS, Professor of RAdiology, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20884/25-8-11
Record Dates: First submitted 2011-12-02; First posted 2012-01-25 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Arterial Occlusive Disease
Keywords: Drug coated balloons; Drug eluting stents
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug Coated Balloon (DCB) Arm (Experimental): Patients included in this arm will undergo PTA with the use of a paclitaxel coated balloon.
  Interventions: Procedure: Paclitaxel coated balloon angioplasty.
- Drug Eluting Stents (DES) Arm (Active Comparator): Patients in this arm will undergo primary infrapopliteal stenting of the target lesion using a drug-eluting stent.
  Interventions: Procedure: Infrapopliteal Primary Drug Eluting Stenting

INTERVENTIONS:
Procedure: Paclitaxel coated balloon angioplasty. — Infrapopliteal angioplasty using a paclitaxel coated balloon.
  Other Names: DCB
  Arms: Drug Coated Balloon (DCB) Arm
Procedure: Infrapopliteal Primary Drug Eluting Stenting — Infrapopliteal primary stenting using drug-eluting stent(s)
  Other Names: DES
  Arms: Drug Eluting Stents (DES) Arm

SUMMARY:
In total 50 patients diagnosed with long-segment infrapopliteal arterial disease will be randomized in two groups. The patients randomized in the Drug coated balloons (DCB) study arm will undergo a percutaneous transluminal angioplasty (PTA) with the use of a paclitaxel-coated balloon, while the patients randomized in the drug-eluting stent (DES) study arm will undergo primary stenting using drug-eluting stent(s). The study's primary endpoints will be the 6-month angiographic binary restenosis rate. Secondary endpoints will include the immediate technical success,6-month primary patency, target lesion revascularization and limb salvage and complication rates.

DETAILED DESCRIPTION:
Patients programmed to undergo PTA due to angiographically-proven infrapopliteal arterial disease in our department will be randomized in the above mentioned study arms. The studies primary endpoint will be assessed with the use of intra-arterial digital subtracted angiography and subsequent Quantitative Vascular Analysis (QVA) analysis.Clinical follow-up is set at 1, 3 and 6 months. Patients' baseline demographics and procedural details will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Angiographically documented infrapopliteal disease.
* Rutherford category of peripheral arterial disease between class 3 to 6
* Lesion length between 70 to 220 mm
* Lesions situated in the proximal, mid and mid to distal segments of the tibial vessels.

Exclusion Criteria:

* Lesion length < 70 mm or > 220 mm.
* Lesions situated in the distal third of the tibial vessels

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Angiographic Binary Restenosis | 6 months
  Angiographic binary restenosis of the target lesion defined by quantitative vessel analysis at 6 months follow-up

SECONDARY OUTCOMES:
Technical success rate | intra-procedural
  Successful balloon angioplasty without stent use due to flow limiting dissection or/and <30% remaining target lesion stenosis in the DCB arm and successful balloon angioplasty without flow limiting dissection or/and <30% remaining target lesion stenosis in the DES arm.
Procedure related complication rates | up to 30 days
  procedure related major and minor complication rates identified during the procedure or within 30 days after the completion of the procedure.
Target lesion revascularization | 6 months
  Clinically-driven target lesion re-intervention
Limb salvage | 6 months
  Major amputation-free interval of the treated limb at 6 months follow-up
Angiographic Primary Patency | 6 months
  Angiographically proven target lesion patency without any additional revascularization procedure

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Siablis, MD,PhD, Study Chair — University Hospital of Patras; Dimitrios Karnabatidis, MD, PhD, Study Director — University Hospital of Patras; Konstantinos Katsanos, MD, PhD, Principal Investigator — University Hospital of Patras; Stavros Spiliopoulos, MD, PhD, Principal Investigator — University Hospital of Patras; Athanasios Diamantopoulos, MD, Principal Investigator — Patras Univesrity Hospital; Panagiotis Kitrou, MD, Principal Investigator — University Hospital of Patras
Locations (1):
- Patras University Hospital, Rio, Achaia, Greece

REFERENCES:
- [Derived] Siablis D, Kitrou PM, Spiliopoulos S, Katsanos K, Karnabatidis D. Paclitaxel-coated balloon angioplasty versus drug-eluting stenting for the treatment of infrapopliteal long-segment arterial occlusive disease: the IDEAS randomized controlled trial. JACC Cardiovasc Interv. 2014 Sep;7(9):1048-56. doi: 10.1016/j.jcin.2014.04.015. PMID 25234679